CLINICAL TRIAL: NCT07011095
Title: A Pilot Trial to Assess the Feasibility of a Multicentre, Phase IV, Prospective, Randomized, Open-label, Two-arm Study With Blinded-endpoint Evaluation to Investigate Vitamin K Antagonist (VKA) Therapy Compared With Direct Oral Anticoagulant (DOAC) Therapy in Male and Female Participants With Atrial Fibrillation and Recent Ischemic Stroke While on a DOAC
Brief Title: DOAC or VKA in Patients With AF and Stroke While on DOAC - a Pilot Trial
Acronym: SWITCH-AF
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SWITCH-AF - Pilot
Record Dates: First submitted 2025-05-27; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation (AF); Stroke (in Patients With Atrial Fibrillation)
Keywords: stroke; atrial fibrillation; A-Fib; SWITCH-AF; DOAC; Warfarin; Anticoagulant
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — N(4)-oleylcytosine arabinoside; Rivaroxaban; Dabigatran; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VKA Arm (Experimental): Vitamin K Antagonist
  Interventions: Drug: VKA
- DOAC Arm (Experimental): Direct oral anticoagulant (locally approved)
  Interventions: Drug: Direct Oral Anticoagulant (DOAC)

INTERVENTIONS:
Drug: VKA — Warfarin
  Arms: VKA Arm
Drug: Direct Oral Anticoagulant (DOAC) — Locally approved DOACs
  Other Names: Rivaroxaban (Xarelto); Dabigatran (Pradaxa); Apixaban (Eliquis)
  Arms: DOAC Arm

SUMMARY:
People with atrial fibrillation who have a stroke while receiving a DOAC are at increased risk of experiencing another stroke. Physicians do not know the best medication to prevent another stroke in this group of people. Options include continuing the same DOAC, switching to another DOAC or switching to warfarin.

The investigators of the SWITCH-AF trial are trying to find out whether switching to warfarin or continuing a DOAC is better for preventing stroke.

The purpose of this study, called a pilot study, is to test the study plan and to find out whether enough participants will join a larger study that answers the question. A pilot study involves a small number of participants and it is not expected to tell us which treatment is better.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided.
2. Age >18 years.
3. Documented history of AF or atrial flutter.
4. Ischemic stroke while on a DOAC within 14 days prior to enrollment identified on imaging.
5. In the opinion of the investigator, it is safe to initiate oral anticoagulation with either a VKA or a DOAC within 24 hours of randomization-

Exclusion Criteria:

1. There is strong evidence for the qualifying stroke event to be associated with permanent discontinuation of DOAC therapy (for any reason)
2. Patient is unable or unwilling to take oral anticoagulation
3. History of intracranial bleeding.
4. Patient is on chronic hemodialysis or likely to need renal replacement therapy during the course of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-03 (Estimated); Primary Completion 2027-02-03 (Estimated); Study Completion 2027-06-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment | From site activation until the end of recruitment (approximately 24 months)
  Recruitment rate; 1 patient per month per center at 9 Canadian stroke centers

SECONDARY OUTCOMES:
Feasibility - Adherence to Assigned Medication | Enrollment to final visit (average 12 months)
  Proportion of participants who cross-over (i.e., vitamin K antagonist to DOAC, or DOAC to vitamin K antagonist) is <5%
Feasibility - Retention | At 6 months from randomization
  Retention of ≥95% of study participants